CLINICAL TRIAL: NCT06640751
Title: The Effect of Interventions for Health Behaviors in Hypertensive Patients -Based on the PRECEDE-PROCEED Model
Brief Title: The Effect of Interventions for Health Behaviors in Hypertensive Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yuan He, Prof., Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2021378
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Hypertension; Health Behavior; Public Health
MeSH Terms: conditions — Hypertension; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group, based on the three core elements of the PROCEED model (predisposing, enabling, and reinforcing factors), aims to influence the health behaviors of patients with hypertension.
  Interventions: Behavioral: Health behavior intervention
- Control (No Intervention): During the study, control participant will be provided with existing community health education on hypertension.

INTERVENTIONS:
Behavioral: Health behavior intervention — The program is a group-based intervention provided by a healthcare team consisting of researchers, cardiologists, family doctors, community healthcare workers, psychologists, and health education specialists. The intervention is structured around three modules-predisposing, enabling, and reinforcing factors-that provide a framework for educational interventions aimed at promoting healthy behaviors in hypertensive patients.
  Arms: Intervention

SUMMARY:
Hypertension is a major risk factor for cardiovascular disease, chronic kidney disease, and premature death worldwide. With an aging population and changes in dietary patterns and lifestyles, the prevalence of hypertension is rising globally, especially in developing countries. Hypertension is the most common chronic disease and a growing public health problem in China. A recent study estimated the prevalence of hypertension to be 28.56 % ± 10.44 %, ranging from 14.28% to 44.28% among the Chinese population aged over 15 years. The PRECEED-PROCEDE model provides a framework to help health planners and policymakers design effective health interventions based on evaluation and analysis of situations. This model has been used in different recent studies related to behavioral change. The study aims to examine the effectiveness of interventions for health behaviors in hypertensive patients based on the PRECEDE-PROCEED model.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with mild to moderate primary hypertension according to the diagnostic criteria of the "2018 Revised Edition of the Chinese Guidelines for the Prevention and Treatment of Hypertension," whose blood pressure is not well controlled or who have poor treatment compliance;
2. Age greater than 18 years and less than 80 years;
3. Normal language communication ability and willingness to participate in the study;
4. Have lived in the community for at least 12 months.

Exclusion Criteria:

1. Patients who lack basic behavioral abilities, have impaired memory function, or have limited language expression abilities;
2. Patients who are simultaneously participating in other intervention studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Health behavior | 1. Before the intervention: Baseline 2. During the intervention (at the end of the 3th, 6th month of the study) 3. the follow-up test (posttests - at the end of the 9th month of the study)
  Health behaviors associated with hypertensive patients, including treatment adherence, physical activity. Treatment adherence will be measured by the Chinese version of Hill-Bone compliance to high blood pressure therapy scale (HBTS). Each item is rated on a 4-point Likert scale, ranging from 1 (All the Time) to 4 (None of the Time), with a higher score reflecting a better outcome. Physical activity will be measured by the International Physical Activity Questionnaire-Short Form (IPAQ-SF). The IPAQ-SF is a self-administered questionnaire, which is used to measure individuals' physical activity during the last seven days. Participants were required to report the frequency and duration that they engaged in each intensity activity. The total score is the summation of the duration and frequency of walking, moderate-, and vigorous-intensity activities, which was reported as the "metabolic equivalent of task-min per week. This instrument has been widely used and well validated.
systolic blood pressure | 1. Before the intervention: Baseline 2. During the intervention (at the end of the 3th, 6th month of the study) 3. the follow-up test (posttests - at the end of the 9th month of the study)
  change in SBP between the intervention and control at 9 months
Delay discounting | 1. Before the intervention: Baseline 2. During the intervention (at the end of the 3th, 6th month of the study) 3. the follow-up test (posttests - at the end of the 9th month of the study)
  Self-written computer program. Discount rates from the delay discounting task were calculated with hyperbolic discounting model of the form: V= A/(1+kD). A higher value of k value indicates a greater discount for delayed rewards.

SECONDARY OUTCOMES:
Knowledge of hypertension | 1. Before the intervention: Baseline 2. During the intervention (at the end of the 3th, 6th month of the study) 3. the follow-up test (posttests - at the end of the 9th month of the study)
  Self-compiled questionnaire. It consisted of 16 binary items. A score of 1 was given for each correct answer, and a score of 0 was given for incorrect and "don't know" replies for each question, with a higher score reflecting a better outcome.
Reinforcing factors | 1. Before the intervention: Baseline 2. During the intervention (at the end of the 6th month of the study) 3. the follow-up test (posttests - at the end of the 9th month)
  The questionnaire of reinforcing factors will be designed based on the precede - proceed model. Each item is rated on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree), with a higher score reflecting a better outcome.
Enabling factors | 1. Before the intervention: Baseline 2. During the intervention (at the end of the 6th month of the study) 3. the follow-up test (posttests - at the end of the 9th month)
  The questionnaire of enabling factors will be designed based on the precede - proceed model. Each item is rated on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree), with a higher score reflecting a better outcome.
Self-efficacy | 1. Before the intervention: Baseline 2. During the intervention (at the end of the 3th, 6th month of the study) 3. the follow-up test (posttests - at the end of the 9th month)
  the Chinese version of the Perceived Health Competence Scale (PHCS). Each item is rated on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5(strongly agree), with a higher score reflecting a better outcome. This instrument has been widely used and well validated.

CONTACTS AND LOCATIONS:
Locations (1):
- Community health service center, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No